CLINICAL TRIAL: NCT06151717
Title: PRAGMMATIC: A Comparative Clinical Trial to Determine the BEST Initial Therapy for Multiple Myeloma
Brief Title: A Comparative Clinical Study to Determine the Optimal Initial Therapy for Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC230811; NCI-2023-09520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC230811 (Other: Mayo Clinic); PRAGMMATIC (Other: Mayo Clinic); 23-006335 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the outcomes of patients undergoing initial therapy for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the overall survival between bortezomib, lenalidomide and dexamethasone (VRd), daratumumab, lenalidomide and dexamethasone (DRd) and daratumumab, bortezomib, lenalidomide and dexamethasone (DVRd) used as initial therapy for patients with newly diagnosed MM.

OUTLINE: This is an observational study.

Patients have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated active multiple myeloma starting a new treatment for the disease with one of the three established treatment regimens: VRd (bortezomib, lenalidomide, dexamethasone), DRd (daratumumab lenalidomide dexamethasone), or DVRd (daratumumab, bortezomib, lenalidomide, and dexamethasone)
* No prior treatment for myeloma
* Not receiving concurrent treatment for another active malignancy
* No more than 3 months from start of treatment

Exclusion Criteria:

* Does not meet all inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with previously untreated multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | Every 3 months, up to 10 years
  Overall survival, defined as the time from initiation of therapy to the time of death due to any cause, will be assessed by review of medical record, contacting the participant, or contacting the participant's local physician every 3 months for up to 10 years after participant starts the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials